CLINICAL TRIAL: NCT00969215
Title: Burn Scar Characteristics After Treatment With Fractional CO2 Laser: A Clinical and Histological Study
Brief Title: Burn Scar Appearance After Treatment With Fractional Carbon Dioxide (CO2) Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moy-Fincher Medical Group (Other)
Responsible Party: Ronald Moy, MD, Moy-Fincher Medical Group
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MF-02
Record Dates: First submitted 2009-08-29; First posted 2009-09-01 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Scars
Keywords: burn scar; fractional carbon dioxide laser; scar revision
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser treatment (Experimental): Half of each subject's scar will be treated with a fractional CO2 laser.
  Interventions: Device: Lumenis fractional carbon dioxide laser
- No treatment (No Intervention): Half of each subject's scar will not be treated.

INTERVENTIONS:
Device: Lumenis fractional carbon dioxide laser — Laser resurfacing of a burn scar
  Other Names: Lumenis
  Arms: Laser treatment

SUMMARY:
The purpose of this study is to determine if fractional carbon dioxide laser treatment of a burn scar is a more effective method for improving the appearance of scars than the current available treatments.

ELIGIBILITY:
Inclusion Criteria:

* Have a mature burn scar and desire revision
* Fluent in English
* Must reside in the Los Angeles vicinity for the duration of the study

Exclusion Criteria:

* Previous history of scar revision
* Non-English speakers
* Pregnant or cognitively impaired subjects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Evidence of clinical improvement of burn scar appearance as determined by blinded-observer and patient ratings. | 2 weeks after each procedure

CONTACTS AND LOCATIONS:
Overall Officials: David Ozog, MD, Principal Investigator — Moy-Fincher Medical Group
Locations (1):
- Moy-Fincher Medical Group, Los Angeles, California, United States